CLINICAL TRIAL: NCT01472744
Title: Influence of Fitness on Brain and Cognition II
Brief Title: Fit & Active Seniors Trial
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Edward McAuley, Professor, Kinesiology and Community Health, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R37AG025667 (NIH); 392 (Other Grant/Funding Number: Center for Nutrition, Learning and Memory UIUC)
Record Dates: First submitted 2011-08-18; First posted 2011-11-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Aging
Keywords: Executive function; Aging; Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Walking; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dance (Experimental): Participants will be instructed in various forms of dances such as ballroom, swing, waltz, folk, and English country.
  Interventions: Behavioral: Dance Group
- Strengthening, Stability, Stretching (Active Comparator): Participants will be instructed in various forms of strength, stretching (flexibility) and stability (balance)exercises.
  Interventions: Behavioral: Strength, Stretching, Stability
- Walking (Experimental): Participants in this moderate aerobic conditioning exercise program will be instructed in a walking program that focuses on having them walk within their target heart rate.
  Interventions: Behavioral: Walking
- Walking + Nutritional Supplement (Experimental): Participants in this moderate aerobic conditioning exercise program will be instructed in a walking program that focuses on having them walk within their target heart rate. These participants will also be provided with a daily nutritionally balanced liquid, milk-based formula.
  Interventions: Behavioral: Walking; Behavioral: Walking + Nutrition

INTERVENTIONS:
Behavioral: Dance Group — Participants will be instructed and learn various forms of dance (i.e. English country, folk, ballroom) and will be led by trained dance instructors and exercise specialists. Participants will for one-hour sessions and meet three times per week for six months.
  Other Names: Fit & Active Seniors Trial
  Arms: Dance
Behavioral: Strength, Stretching, Stability — Exercises focusing on strength, flexibility and balance will be performed at one-hour sessions held three times per week for six months. Classes are led by trained exercise specialists.
  Other Names: Fit & Active Seniors Trial
  Arms: Strengthening, Stability, Stretching
Behavioral: Walking — Participants in this moderate aerobic conditioning exercise program will be instructed in a walking program that focuses on having them walk within their target heart rate. They will be provided with heart rate monitors and pedometers for accurate record keeping. They will meet three times per week for one hour for six months. Warm up and cool down stretches will be a part of each walking session and sessions will be monitored and led by trained exercise specialists.
  Arms: Walking; Walking + Nutritional Supplement
Behavioral: Walking + Nutrition — Participants in this moderate aerobic conditioning exercise program will be instructed in a walking program that focuses on having them walk within their target heart rate. They will be provided with heart rate monitors and pedometers for accurate record keeping. They will meet three times per week for one hour for six months. Warm up and cool down stretches will be a part of each walking session and sessions will be monitored and led by trained exercise specialists. These participants will also be provided with a daily nutritionally balanced liquid, milk-based supplement formula.
  Arms: Walking + Nutritional Supplement

SUMMARY:
The investigators propose to test the hypothesis that a six-month intervention of combined fitness and cognitive training in the form of dancing will have a significant positive effect on a variety of executive control and memory processes as well as brain structure and function as compared to a non-aerobic strength and balance control/comparison group. Additionally, these two groups will be compared to walking groups in which one of the walking groups will also be provided with a daily, liquid, milk-based nutritional supplement.

DETAILED DESCRIPTION:
Our previous trial (known as HALT, Healthy Active Lifestyle Trial) suggests that improvements in aerobic fitness have beneficial effects on cognitive function that are rather specific. That is, improvements in aerobic fitness appear to result in improvements in executive control processes such as scheduling, planning, coordination, inhibition, and working memory - some of the very cognitive abilities most affected during aging. Indeed, executive control processes and the prefrontal and frontal regions which support them have shown substantial and disproportionate age-related declines. The main hypothesis that the investigators test in the present project is that such deficits may be particularly benefited by improvements in aerobic fitness combined with cognitive training in the form of dance. Additionally, we will compare the outcomes of these interventions with an aerobic condition (walking) group and an aerobic condition (walking) group that also is provided with a daily nutritional supplement (walking + nutrition). The investigators will examine the relationship between aerobic fitness, physical activity, cognitive status, and brain function with this six-month aerobic training intervention study. The investigators will collect psychosocial data and functional fitness data to assess other relevant changes in psychological and physical function brought about by exercise training. Healthy, non-active older adults (60 to 79 years of age) will be recruited from the local community. Half One quarter of the older adults will be randomly assigned to an aerobic/cognitive combination group (dance), one quarter will be while the remaining half of the older adults will be randomly assigned to a non-aerobic control group (stretching, strengthening, and stability), one quarter will be assigned to the walking group, and one quarter will be assigned to the walking + nutrition group. The exercise interventions will be conducted by trained exercise staff. The participants will be assessed before and after the intervention (6 months). Assessments will include (a) cardiorespiratory testing, (b) physical activity monitoring (c) performance on neurocognitive tests of executive and non-executive function (d) measures of brain activation (fMRI) during cognitive tasks in a 3.0 tesla MRI system (e) a battery of psychosocial questionnaires (f) functional performance measures and (g) a mock street walking task.

ELIGIBILITY:
Inclusion Criteria:

* 60-79 years of age
* Low-active: zero to two days of physical activity (> 30 minutes per day) per week in previous six months.
* Personal physician's examination and/or consent to participate in testing and exercise intervention
* Successful completion of graded exercise test without evidence of cardiac abnormalities or responses which are likely to be exacerbated by exercise. This decision will be made by the attending cardiologist.
* Adequate responses to the Telephone Interview of Cognitive Status (TICS-M) questionnaire
* Corrected (near and far) acuity of 20/40 or better in both eyes and no diagnosis of color-blindedness
* Initial depression score on GDS-15 (Geriatric Depression Scale) below clinical level (> 10)
* No presence of implanted devices or metallic bodies above the waist
* No history of brain surgery that involved removal of brain tissue
* Right-handed
* No history of stroke or Transient ischemic attack(TIA)
* Intention to remain in the local area for the duration of the intervention or testing period
* English fluency

Exclusion Criteria:

* Below 60 years of age or above 80 years of age at beginning of intervention
* Self-reported regular physical activity of more than 2 times per week in last six months
* Non-consent of physician
* Evidence of abnormal cardiac responses or conditions during graded exercise testing
* Inadequate responses to the Telephone Interview of Cognitive Status (TICS-M) questionnaire (<20)
* Uncorrectable (near and far) acuity of greater than 20/40 in either eye and/or color-blindness
* Depression score on GDS-15 indicative of clinical depression (≤ 10)
* Presence of any implanted devices above the waist i.e. cardiac pacemaker or auto-defibrillators; neural pacemaker; aneurysm clips in the Central Nervous System(CNS); cochlear implant; metallic bodies in the eye or CNS; any form of wires or metal devices that may concentrate radiofrequency fields
* History of brain surgery that involved removal of brain tissue
* Left-handed
* History of Stroke or TIA
* Intent to move or be away from the area for an extended period of time (i.e. > 3 weeks) during the intervention or testing period
* Inability to communicate effectively in English

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to month six in brain structure and function | Baseline and six months
  Participants will undergo a neuropsychological battery of tasks assessing memory, attention and decision-making at baseline and month six. They will also undergo an fMRI during which images of brain structure and function (completing tasks during image collection) will be compared from baseline to month six.
Change from baseline to month six in cardiorespiratory fitness | Baseline and six months
  We will conduct graded maximal exercise treadmill test measuring peak oxygen consumption at baseline and six months.

SECONDARY OUTCOMES:
Change from baseline to month six: Quality of life | Baseline and six months
  We will assess multiple indicators of Quality of Life such as: depression; physical and mental health status; satisfaction with life; etc.
Change from baseline to month six: Self-efficacy | Baseline, three weeks and six months
  We will examine the extent to which self-efficacy (e.g. barriers, adherence, function) changes as a function of participation in regular group physical activity training.
Program adherence over six month intervention | Six months
  We will monitor attendance during the six-month intervention(program meets three days per week).
Change from baseline to month six: Physical function | Baseline and six months
  We will conduct functional fitness testing including tests of balance, strength, mobility and flexibility at baseline and six months.
Change from baseline to month six: Psychosocial Outcomes | Baseline and six months
  We will assess changes in psychosocial function (e.g. self-esteem; social support; anxiety) by written questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Kramer, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendez Colmenares A, Voss MW, Fanning J, Salerno EA, Gothe NP, Thomas ML, McAuley E, Kramer AF, Burzynska AZ. White matter plasticity in healthy older adults: The effects of aerobic exercise. Neuroimage. 2021 Oct 1;239:118305. doi: 10.1016/j.neuroimage.2021.118305. Epub 2021 Jun 24. PMID 34174392
- [Derived] Burzynska AZ, Voss MW, Fanning J, Salerno EA, Gothe NP, McAuley E, Kramer AF. Sensor-measured sedentariness and physical activity are differentially related to fluid and crystallized abilities in aging. Psychol Aging. 2020 Dec;35(8):1154-1169. doi: 10.1037/pag0000580. Epub 2020 Sep 24. PMID 32969693
- [Derived] Gothe NP, Ehlers DK, Salerno EA, Fanning J, Kramer AF, McAuley E. Physical Activity, Sleep and Quality of Life in Older Adults: Influence of Physical, Mental and Social Well-being. Behav Sleep Med. 2020 Nov-Dec;18(6):797-808. doi: 10.1080/15402002.2019.1690493. Epub 2019 Nov 12. PMID 31713442
- [Derived] Baniqued PL, Gallen CL, Voss MW, Burzynska AZ, Wong CN, Cooke GE, Duffy K, Fanning J, Ehlers DK, Salerno EA, Aguinaga S, McAuley E, Kramer AF, D'Esposito M. Brain Network Modularity Predicts Exercise-Related Executive Function Gains in Older Adults. Front Aging Neurosci. 2018 Jan 4;9:426. doi: 10.3389/fnagi.2017.00426. eCollection 2017. PMID 29354050
- [Derived] Awick EA, Ehlers DK, Aguinaga S, Daugherty AM, Kramer AF, McAuley E. Effects of a randomized exercise trial on physical activity, psychological distress and quality of life in older adults. Gen Hosp Psychiatry. 2017 Nov;49:44-50. doi: 10.1016/j.genhosppsych.2017.06.005. Epub 2017 Jun 15. PMID 28662897
- [Derived] Ehlers DK, Daugherty AM, Burzynska AZ, Fanning J, Awick EA, Chaddock-Heyman L, Kramer AF, McAuley E. Regional Brain Volumes Moderate, but Do Not Mediate, the Effects of Group-Based Exercise Training on Reductions in Loneliness in Older Adults. Front Aging Neurosci. 2017 Apr 25;9:110. doi: 10.3389/fnagi.2017.00110. eCollection 2017. PMID 28487648
- [Derived] Burzynska AZ, Jiao Y, Knecht AM, Fanning J, Awick EA, Chen T, Gothe N, Voss MW, McAuley E, Kramer AF. White Matter Integrity Declined Over 6-Months, but Dance Intervention Improved Integrity of the Fornix of Older Adults. Front Aging Neurosci. 2017 Mar 16;9:59. doi: 10.3389/fnagi.2017.00059. eCollection 2017. PMID 28360853
- [Derived] Ehlers DK, Banducci SE, Daugherty AM, Fanning J, Awick EA, Porter GC, Burzynska A, Shen S, Kramer AF, McAuley E. Effects of Gait Self-Efficacy and Lower-Extremity Physical Function on Dual-Task Performance in Older Adults. Biomed Res Int. 2017;2017:8570960. doi: 10.1155/2017/8570960. Epub 2017 Feb 1. PMID 28255557
- [Derived] Ehlers DK, Fanning J, Awick EA, Kramer AF, McAuley E. Contamination by an Active Control Condition in a Randomized Exercise Trial. PLoS One. 2016 Oct 10;11(10):e0164246. doi: 10.1371/journal.pone.0164246. eCollection 2016. PMID 27723781
- See also: Exercise Psychology Laboratory — http://epl.illinois.edu